CLINICAL TRIAL: NCT00087542
Title: Treatment of Hallucinosis/Psychosis in Parkinson's Disease by an Investigational Drug
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: ACP-103-006
Record Dates: First submitted 2004-07-09; First posted 2004-07-14 (Estimated); Last update posted 2005-12-07 (Estimated); Status verified 2005-12

CONDITIONS: Hallucinations; Psychoses; Parkinson's Disease
Keywords: Hallucinosis/Psychosis
MeSH Terms: conditions — Hallucinations; Psychotic Disorders; Parkinson Disease | interventions — pimavanserin

INTERVENTIONS:
Drug: ACP-103

SUMMARY:
The primary objective is to demonstrate that the investigational new drug, ACP-103, is well tolerated by, and will not worsen parkinsonism in, patients with Parkinson's disease and psychosis. The secondary objectives are to determine whether ACP-103 will ameliorate psychosis in patients with Parkinson's disease and whether ACP-103 is safe in Parkinson's disease patients taking multiple anti-parkinsonian medications.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, randomized, placebo-controlled, double-blind trial of four weeks of ACP-103 treatment of psychosis in Parkinson's disease, with four weeks follow-up.

A total of 60 patients meeting entrance criteria will be randomly assigned to receive placebo (30 patients) or active drug (30 patients). Subjects will take study drug daily starting on Day 1. Dose escalations can occur on Study Days 8 and 15 only, and patients will receive a stable daily dosage from Day 16 until Day 28. Single step dose reductions are allowed during that period for adverse events or intolerance.

Patients will be evaluated at screening/baseline and at Study Days 1, 8, 15, 28, and 57 by raters blinded to the treatment. The major response variable will be motoric tolerability. Secondary response variables will be efficacy against psychosis and safety.

Currently, there are no approved drugs for this indication in the United States. Psychotic symptoms in Parkinson's disease patients are almost always stable, often non-threatening, and rarely paranoid or violent in content. The trial includes the requirement that each patient enrolled has a reliable caretaker who will accompany the patient to each visit who can reliably report on the patient's daily level of function. These factors argue for the safe inclusion of a four-week period of placebo treatment.

ELIGIBILITY:
Inclusion Criteria

Male and female patients of any ethnic group and of any age are eligible for participation in this study, providing they meet all the following criteria:

* Subjects with a clinical diagnosis of idiopathic Parkinson's disease, defined as the presence of at least three of the cardinal features of the disease including: rest tremor, rigidity, bradykinesia and/or akinesia, postural balance abnormalities, in the absence of alternative explanations or atypical features.
* Psychosis, defined by the presence of visual and/or auditory hallucinations, with or without delusions, of at least four weeks duration.
* Psychosis, assessed by items A and B of the NPI, and defined as Hallucinations (Frequency x Severity) and Delusions (Frequency x Severity) = a total score of 4 or greater.
* Stable anti-Parkinsonian medication(s) use for at least one week prior to study entry.
* A reliable caretaker who will accompany the subject to each visit, and who can reliably report on the subject's daily level of function.

Exclusion Criteria

Patients who meet any of the following conditions are excluded from the clinical study:

* Inability of subject or caretaker to provide informed consent.
* Pregnant or breastfeeding. Female subjects of child-bearing potential must have a negative urine pregnancy test at screening.
* Female subjects must be of non-childbearing potential or must comply with double-barrier protection methods against conception during the study and for at least one month prior to randomization and one month following completion of the study.
* Presence of any systemic factor contributing to the psychosis such as urinary infection, liver disease, renal failure, anemia, infection, etc. as defined by a comprehensive medical evaluation.
* History of a significant pre-morbid psychiatric condition before the diagnosis of Parkinson's disease, including major depression, mania, or psychotic depression.
* Dementia precluding accurate assessment on psychiatric assessment battery and defined as a score on the MMSE < 21.
* Use of depot neuroleptic within the past year.
* Prior exposure to non-depot neuroleptics within the past 90 days, except for quetiapine or clozapine. Quetiapine and clozapine-treated patients may be enrolled if these agents were discontinued due to drug intolerability. Such patients must not have taken these drugs within the past two weeks.
* Use of the following drugs within the past two weeks: benztropine, biperiden, trihexylphenidyl, amitriptyline, clomipramine, desipramine, nortriptyline, imipramine, doxepin, fluvoxamine, mirtazepine, nefazodone and trazodone.
* Change of anti-depressant, anxiolytic, anticholinergic (specifically oxybutynin, tolterodine), or cognitive enhancer (specifically rivastigmine, tacrine, donepezil, galantamine) dose within the past 30 days and during the 28-day duration of the trial.
* Use of any investigational product within the past 30 days.
* Inability to tolerate a stable level of anti-parkinsonian medications for one week.
* Uncontrolled angina or history of a myocardial infarction within the past three months.
* Concurrent illness that would make use of ACP-103 potentially hazardous.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2004-03; Study Completion 2005-12

PRIMARY OUTCOMES:
ACP-103 is an effective treatment for Parkinson's Disease with psychosis

SECONDARY OUTCOMES:
ACP-103 does not cause worsening of motor function in Parkinson's Disease

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Fountain Valley, California
  - Sunnyvale, California
  - Danbury, Connecticut
  - Pompano Beach, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Kansas City, Kansas
  - Elkridge, Maryland
  - Albany, New York
  - Asheville, North Carolina
  - Philadelphia, Pennsylvania
  - Pawtucket, Rhode Island
  - Brentwood, Tennessee